CLINICAL TRIAL: NCT04023617
Title: A Study of Nivolumab +/- Docetaxel in Patients Previously Treated With Advanced or Metastatic Non Small Cell Lung Cancer
Brief Title: A Study of Nivolumab +/- Docetaxel in Patients Previously Treated With Advanced or Metastatic NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jian Fang, Department of Thoracic Oncology II, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDO-101
Record Dates: First submitted 2019-07-08; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Docetaxel; Nivolumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivolumab + Docetaxel (Experimental): Nivolumab was administered at a dose of 300 mg on the first day of the 21-day cycle (every 3 weeks; q3w) when combined with docetaxel, and administered at a dose of 200 mg on the first day of each 14-day cycle (every 2 weeks; q2w) after stopping docetaxel treatment.
  On the first day of each cycle (21 days), docetaxel 75 mg/m2 was infused by IV on Day 1 of each 21-day cycle for 4-6 cycles (judged by investigator).
  Interventions: Drug: Nivolumab
- Nivolumab (Active Comparator): Nivolumab was administered in the monotherapy group at a dose of 200 mg on the first day of each 14-day cycle (every 2 weeks; q2w).
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 300mg + docetaxel 75mg/m2 IV q3w Nivolumab 200mg IV q2w
  Other Names: docetaxel

SUMMARY:
This study is a randomized, single-center, open-label, phase II clinical trial designed to evaluate non-small cell lung cancer that has failed to undergo excessive platinum-based chemotherapy and has not received excessive statin chemotherapy and has not received immunotherapy. The efficacy and safety of Nivolumab in combination with docetaxel and Nivolumab in patients.

Qualified patients were stratified by histological type (squamous cell carcinoma vs. non-squamous cell carcinoma) randomized to receive the following regimen in a 1:1 ratio:

Group A: Nivolumab 300mg + docetaxel 75mg/m2 IV q3w Group B: Nivolumab 200mg IV q2w All patients were evaluated for tumor at baseline, and tumor evaluations were performed every 6 weeks within 48 weeks after randomization (regardless of whether dosing was delayed). After the 48th week of assessment, a tumor assessment is required every 9 weeks until disease progression, withdrawal of informed consent, sponsor termination study, or patient death.

DETAILED DESCRIPTION:
Nivolumab and Docetaxel have been approved as standard second-line treatments for non-small cell lung cancer in several countries including China and the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Men & women ≥18, and ≤75 years of age.
2. Subjects with histologically or cytologically-documented non-squamous cell NSCLC who present with Stage IIIB/IV disease or recurrent or progressive disease following multimodal therapy (radiation therapy, surgical resection, or definitive chemoradiation therapy for locally advanced disease) and who will receive study therapy as second line of treatment for advanced disease.
3. The patient's tumor must be free of EGFR gene-sensitive mutations (including but not limited to exon 19 deletion mutation or exon 21 L858R mutation, exon 21 L861Q, exon 18 G719X or exon 20 S768I site Mutation) and ALK gene rearrangement. If the pathology is squamous cell carcinoma or the tumor of a known patient has a KRAS mutation, then EGFR and ALK are not required to be detected.
4. Disease recurrence or progression during/after one prior platinum doublet-based chemotherapy regimen for advanced or metastatic disease.
5. Measurable disease by Computed tomography (CT)/Magnetic resonance imaging (MRI) per RECIST 1.1 criteria.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
7. Expected survival time ≥ 12 weeks.
8. Has adequate organ and bone marrow function, defined as follows:

   * Hemoglobin ≥ 9.0 g/dL.
   * Absolute neutrophil count ≥1.5 × 109 /L.
   * Platelet count ≥80 × 109 /L.
   * Serum total bilirubin ≤ 1.5 × normal upper limit (ULN); for patients with liver metastasis, serum total bilirubin ≤ 5 × normal upper limit (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; for patients with liver metastases: ALT and AST ≤ 5 × ULN.
   * Serum creatinine (Cr) ≤ 1.5 times the upper limit of normal (ULN).
9. Pre-menopausal women have a negative urine or serum pregnancy test within 14 days prior to initiation of treatment.
10. Written informed consent was signed prior to the experiment.

Exclusion Criteria:

1. Have been treated with docetaxel or have previously received immunological checkpoint inhibitors targeting PD-1, PD-L1 or CTLA-4.
2. Prior to randomization ≤ 21 days (or ≤ 5 half-lives, whichever is shorter) have received chemotherapy, other test drugs, and Chinese herbal medicines used to control cancer.
3. Uncontrolled brain metastases and all meningeal metastases. Stereotactic radiotherapy within 7 days prior to the start of treatment in the first cycle, or brain metastases who underwent whole brain radiotherapy within the first 14 days (if the patient detected a new asymptomatic CNS metastasis during the screening scan, then radiotherapy must be received) And/or central nervous system metastases. After treatment, these patients do not require additional brain scans to enter the trial if other inclusion criteria are met.
4. Large area radiotherapy (except for local palliative radiotherapy for bones).
5. Pericardial effusion, pleural effusion, or ascites that is clinically uncontrolled and requires pericardial puncture, thoracic puncture, or abdominal puncture drainage within 2 weeks of randomization.
6. A history of malignancy other than NSCLC within the first 5 years of randomization, except for malignant tumors with a very low risk of metastatic death and expected to heal after treatment (eg fully treated cervical carcinoma in situ, basal or squamous cell skin cancer, accepted Localized prostate cancer for radical treatment, ductal carcinoma in situ for radical surgery).
7. Have undergone major surgery (as defined by the investigator) within 28 days prior to the first dose. Note: For the purpose of palliative care, local surgical treatment of isolated lesions is acceptable.
8. Any condition that, depending on the investigator's judgment, interferes with the evaluation of the efficacy of the study drug or explains the patient's safety or findings, including but not limited to: persistent or active infection, symptomatic congestive heart failure, poorly controlled hypertension, Unstable angina, arrhythmia, or psychiatric/social conditions that affect the study's requirements, significantly increase the risk of AEs in the study drug, or affect the patient's ability to provide informed consent.
9. Active or previously documented autoimmune or inflammatory disease (with vitiligo, hypothyroidism (after Hashimoto's syndrome) and stable disease after hormone replacement therapy, no active disease in the past 5 years Patients can be enrolled).
10. Active infections, including tuberculosis, hepatitis B, and hepatitis C.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 24 months
  progression-free survival

SECONDARY OUTCOMES:
OS | 24 months
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China